CLINICAL TRIAL: NCT03902444
Title: AcandiS Stenting of Intracranial STENosis - regisTry
Acronym: ASSISTENT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Acandis GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: ASSISTENT
Record Dates: First submitted 2019-03-27; First posted 2019-04-04 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Intracranial Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Credo® Stent and NeuroSpeed® PTA balloon catheter: Patients treated with Credo® Stent and NeuroSpeed® PTA balloon catheter in the clinical routine
  Interventions: Device: Credo® Stent, NeuroSpeed® PTA balloon catheter

INTERVENTIONS:
Device: Credo® Stent, NeuroSpeed® PTA balloon catheter — a self-expanding stent is used together with a PTA balloon catheter

SUMMARY:
ASSISTENT is designed to collect comprehensive information on technical and clinical safety of the use of Credo® stent together with the NeuroSpeed® PTA balloon catheter in clinical practice in an open registry.

DETAILED DESCRIPTION:
ASSISTENT is subdivided into two components. The first part only requires recording of data acquired in routine clinical practice during the treatment of patients with intracranial stenosis with the self-expandable Credo® stent until discharge. This comprises demographic data, data concerning the qualifying clinical event, limited data on medical history and medication, information about the intervention including technical success and periprocedural complications or events, and information about events and clinical status during the in-hospital treatment until hospital discharge.

The second part of the registry consists of a follow-up visit 30 days after the interventional procedure which will be conducted outside of clinical practice.

ELIGIBILITY:
Inclusion Criteria:

- Treatment with Credo® for symptomatic atherosclerotic intracranial artery stenosis (see product IFU)

Exclusion Criteria:

* There are no specific exclusion criteria (see product IFU)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over 18 with symptomatic intracranial artery stenosis treated with the self-expandable Credo® stent in the participating sites in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Rate of Technical Success | During interventional procedure
  • Technical Success
Number of Patients with Periprocedural Vascular Events | Periprocedural, until 30 days after the interventional procedure
  * Intracranial haemorrhage (symptomatic / asymptomatic)
  * Death
  * TIA in the region of the target vessel
  * Non-disabling ischemic stroke (MRS 0-2) in the region of the target vessel
  * Disabling ischemic stroke (MRS 3-6) in the region of the target vessel
  * TIA outside the region of the target vessel
  * Non-disabling ischemic stroke (MRS 0-2) outside the region of the target vessel
  * Disabling ischemic stroke (MRS 3-6) outside the region of the target vessel
Number of Patients with Cerebrovascular events | At hospital discharge - befor the patient leaves the hospital after the intervention; up to 2 weeks, whichever came first
  * Intracranial haemorrhage (symptomatic / asymptomatic)
  * Death
  * TIA in the region of the target vessel
  * Non-disabling ischemic stroke (MRS 0-2) in the region of the target vessel
  * Disabling ischemic stroke (MRS 3-6) in the region of the target vessel
  * TIA outside the region of the target vessel
  * Non-disabling ischemic stroke (MRS 0-2) outside the region of the target vessel
  * Disabling ischemic stroke (MRS 3-6) outside the region of the target vessel
Number of Patients with Cerebrovascular Events | 30 days after the interventional procedure
  * Intracranial haemorrhage (symptomatic / asymptomatic)
  * Death
  * TIA
  * Non-disabling ischemic stroke (MRS 0-2)
  * Disabling ischemic stroke (MRS 3-6)
  * Interventional re-treatment of the target vessel

SECONDARY OUTCOMES:
Number of Patients with Dissection of the target vessel | During interventional procedure
Number of Patients with Occlusion of the target vessel | 30 days after the interventional procedure
Number of Patients with Myocardial infarction | 30 days after the interventional procedure
Number of Patients with Severe extracranial hemorrhage (requiring surgical treatment or transfusion) | 30 days after the interventional procedure

CONTACTS AND LOCATIONS:
Overall Officials: Götz Thomalla, MD, Principal Investigator — Unversity Medical Center Hamburg-Eppendorf
Locations (16):
- Germany (16):
  - Universitätsklinikum Knappschaftskrankenhaus Bochum, Bochum
  - Uniklinik Köln, Cologne
  - Universitätsklinikum Düsseldorf Institut für Diagnostische und Interventionelle Radiologie Abteilung Neuroradiologie, Düsseldorf
  - Alfried Krupp Krankenhaus Essen, Klinik für Neuroradiologie, Essen
  - Institut für Diagnostische und Interventionelle Neuroradiologie Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Altona, Fachbereich Neuroradiologie, Hamburg
  - Universitätsklinikum Heidelberg Abteilung für Neuroradiologie, Heidelberg
  - Universitätsklinikum Homburg, Homburg
  - Klinikum Ingolstadt, Ingolstadt
  - Otto-von-Guericke-Universität Magdeburg Universitätsklinik für Neuroradiologie, Magdeburg
  - Kliniken Maria Hilf GmbH Mönchengladbach, Klinik für Diagnostische und Interventionelle Radiologie und Neuroradiologie, Mönchengladbach
  - Evangelisches Krankenhaus Oldenburg; Medizinischer Campus Universität Oldenburg, Oldenburg
  - Klinikum Osnabrück, Klinik für Neurologie, Osnabrück
  - KLINIKUM VEST GMBH Knappschaftskrankenhaus Klinik für Radiologie und Neuroradiologie, Recklinghausen
  - St. Lukas Klinik GmbH, radprax MVZ GmbH Solingen, Solingen

IPD SHARING:
Plan to Share IPD: No